CLINICAL TRIAL: NCT02394275
Title: A Prospective Open-Labelled Multi-Centre Trial of Frozen-and-Thawed Fecal Microbiota Transplantation for Recurrent Clostridium Difficile Infection
Brief Title: A Prospective Trial of Frozen-and-Thawed Fecal Microbiota Transplantation for Recurrent Clostridium Difficile Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding for long-term follow-up
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDI.FMT.2
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Clostridium Difficile
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: (Experimental): Eligible patients with receive intervention: frozen fecal microbiota transplantation (FMT), kept at -20 oC and will be thawed prior to administration. Patients on antibiotic to control CDI will discontinue antibiotic 24 hours prior to FMT.
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — All eligible patients will receive fecal microbiota transplant
  Other Names: Human Biotherapy

SUMMARY:
The primary goal of this proposal is to study the outcome of patients with recurrent Clostridium Difficile Infection (CDI) treated with frozen Fecal Microbiota Transplantation (FMT) in an open-labelled controlled trial. The specific objectives are to evaluate the safety of FMT and to determine the clinical response, treatment failure and relapse rate in patients treated with frozen-and-thawed FMT; to assess the functional health and well-being of patients in each arm using the validated tool, and to determine the feasibility of providing standardized FMT in multiple centres across Canada, including community hospitals. The metagenomics will also be conducted from the stool samples collected from select patients from each arm: pre and post treatment and the matching donors. The metagenomics data will be used to determine the bacteria which may have contributed to the cure of CDI.

DETAILED DESCRIPTION:
CDI is the most frequent cause of healthcare-associated infectious diarrhea in industrialized countries and affects over 300,000 patients each year in the United States. The incidence of CDI has nearly tripled between 1996 and 2005 (from 31 to 84 per 100,000 patient-days) in the United States. The rise in incidence has been accompanied by an increase in disease severity, with mortality in up to 6.9% of cases. According to the Canadian Nosocomial Infection Surveillance Program study conducted from November 1, 2004 through April 30, 2005, the incidence rate of health care-associated CDI for adult patients admitted to Canadian hospitals is 65 per 100,000 patient-days. The same study identified that the overall and attributable mortality of patients with CDI is 16.3% and 5.7%, respectively in Canada, which is similar to the US data.1,17 The associated economic burden has also been significant. Nosocomial CDI increases the cost of otherwise matched hospitalizations by four-fold, translating to greater than $1 billion/year (United States). Since the implementation of mandatory reporting of CDI cases in September 2008 in Ontario, more than 13 health-care facilities declared CDI outbreak in Ontario. There were a number of deaths directly due to CDI in these outbreaks. The management of each outbreak is very costly. The direct attributable costs associated with the outbreak management alone per episode per institution exceeded $1 million (direct communication with a hospital chief financial officer).

There is a growing concern regarding failure of standard antimicrobial therapy. The treatment failure rates for metronidazole, which is the ﬁrst line therapy for uncomplicated CDI, have risen from 2.5% to greater than 18% since 2000. Recurrence rates are higher among the elderly, and exceed 50% for those over the age 65.20 Recurrence rates exceed 60% for patients who have failed 3 or more episodes of standard antimicrobial therapies. The vanB gene, which is responsible for conferring vancomycin resistance in Enterococcus has been isolated in clostridia, potentially threatening the future use of vancomycin in CDI.

Given the high failure and recurrence rates using the standard therapy, the principal investigator (PI) of this research proposal has been offering FMT for patients who experienced CDI for longer than 6 months despite multiple courses of metronidazole and oral vancomycin therapy. She began treating patients with recurrent CDI with FMT for the following reasons. First, the patients were not responding to the antibiotic treatment. Second, patients may experience intolerance to metronidazole due to metallic taste, significant nausea and loss of appetite, which can lead to further weight loss as patients with CDI experience considerable weight loss. Also, some patients develop irreversible peripheral neuropathy (nerve damage) with long term use of metronidazole. Third, some of the patients with refractory CDI could not afford to continue with oral vancomycin. The cost of oral vancomycin was prohibitive and they were not routinely reimbursed by the public health plan. A 14-day course of oral vancomycin costs $600 and a number of the patients were on this antibiotic for 6 - 18 months at a cost of $7,200 to $21,600 (personal communication with St. Joseph's Healthcare Outpatient pharmacist). The cost of one FMT is approximately $100, which includes the laboratory screening test and the nurse's administration time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Able to provide informed consent.
3. Laboratory or pathology confirmed diagnosis of recurrent CDI with symptoms (defined below) within the previous 180 days.
4. ≥ 2 episodes of CDI within 6 months and/or ongoing symptoms consistent with CDI despite treatment with oral vancomycin at a dose of at least 125 mg 4 times daily for at least 5 days.

Exclusion Criteria:

1. Planned or actively taking an investigational product for another study.
2. Patients with neutropenia with absolute neutrophil count <0.5 x 109/L
3. Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray
4. Peripheral white blood cell count > 30.0 x 109/L AND temperature > 38.0 oC
5. Active gastroenteritis due to Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia or Campylobacter.
6. Presence of colostomy or ileostomy.
7. Unable to tolerate FMT or enema for any reason.
8. Anticipated requirement for systemic antibiotic therapy for more than 7 days during the 12 week study period.
9. Actively taking Saccharomyces boulardii or probiotics other than yogurt.
10. No symptoms consistent with CDI, off CDI antibiotic therapy for 3 or more weeks
11. Severe underlying disease such that the patient is not expected to survive for at least 30 days.
12. Any condition that, in the opinion of the investigator, that the treatment may pose a health risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants must have laboratory diagnosis of recurrent CDI based on Society for Healthcare Epidemiology of America definition, recurrence defined as return of diarrhea and positive stool test after period of symptom resolution within 8 weeks of the first episode and has received at least 10-day course of oral vancomycin.
  Eligible participants at time of screening will discontinue antibiotic 24 to 48 hours prior to receiving FMT
Period: Overall Study
Arm/Group | Single Arm:
Started | 140
Safety Population | 133
Evaluable at 13 Weeks | 133
Completed | 111
Not Completed | 29
Not completed — Adverse Event | 22
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: 18 years or older with a history of recurrent CDI
Arm/Group | Single Arm:
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (16.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 51
Region of Enrollment [Number; unit: participants]
  Canada | 140

OUTCOME MEASURES:

1. Primary Outcome: No Recurrence of CDI-related Diarrhea
Description: No recurrence of CDI-related diarrhea at 8 weeks following last FMT without the need for an intervention (antibiotics or additional FMT) specifically for recurrence of CDI
Time Frame: 13 weeks
Measure: Number; unit: participants
Groups:
- Single Arm:: Eligible patients with receive intervention: frozen fecal microbiota transplantation (FMT), kept at -20 oC and will be thawed prior to administration.
  Participants on antibiotic to control CDI will discontinue antibiotic 24 - 48 hours hours prior to FMT.
  Fecal Microbiota Transplant: All eligible patients will receive fecal microbiota transplant
Arm/Group | Single Arm:
Number analyzed (Participants) | 133
participants
  FMT open-label | 133
  Treatment Success | 119

2. Secondary Outcome: Safety of FMT
Description: Evaluate safety of FMT for any serious adverse events up to and including week 13 of receiving FMT for any of the following:
  * Death or a life-threatening event
  * Hospitalization or prolongation of current hospitalization
  * A significant new incapacity to conduct normal life functions
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Groups:
- FMT Open-label: Eligible patients received intervention: frozen fecal microbiota transplantation (FMT), kept at -20 oC and thawed prior to administration. Patients on antibiotic to control CDI will discontinue antibiotic 24 hours prior to FMT.
  Fecal Microbiota Transplant: All eligible patients received fecal microbiota transplant
Arm/Group | FMT Open-label
Number analyzed (Participants) | 133
Participants
  All cause mortality | 11
  SAE due to cardiac cause | 4
  SAE due to GI cause | 3
  SAE due to Infections (recurrent C. difficile) | 5
  SAE due to renal cause | 2
  SAE due to respiratory cause | 2

ADVERSE EVENTS:
Arm/Group | Single Arm:
All-Cause Mortality (participants affected / at risk) | 11/133
Serious Adverse Events (participants affected / at risk) | 16/133
Other Adverse Events (participants affected / at risk) | 11/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: (N=133)
Urinary tract infection (Infections and infestations) | 4
Congestive heart failure (Cardiac disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Bacteremia (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: (N=133)
Gastrointestinal disorders (Gastrointestinal disorders) | 11 — abdominal cramps, loose bowel movements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2014-06-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02394275/SAP_000.pdf